CLINICAL TRIAL: NCT02631902
Title: Diabetes em Movimento® - Community-based Lifestyle Intervention Program for Patients With Type 2 Diabetes: Effects on Health and Well-being
Brief Title: Diabetes em Movimento® - Community-based Lifestyle Intervention Program for Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Responsible Party: Principal Investigator, Romeu Duarte Carneiro Mendes, MD, PhD, University of Trás-os-Montes and Alto Douro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTras
Record Dates: First submitted 2015-10-11; First posted 2015-12-16 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes-Related Complications
Keywords: Community-based intervention; Exercise program; Dietary intervention program; Health promotion; Subjective well-being; Cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Exercise; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise (Experimental): Community-based exercise program
  Interventions: Behavioral: Exercise
- Exercise plus dietary intervention (Experimental): Community-based exercise and dietary intervention program
  Interventions: Behavioral: Exercise; Behavioral: Dietary intervention
- Control (No Intervention): Habitual physical activity and habitual dietary pattern

INTERVENTIONS:
Behavioral: Exercise — Community-based exercise program with 3 weekly exercise sessions
  Arms: Exercise; Exercise plus dietary intervention
Behavioral: Dietary intervention — Community-based dietary intervention program
  Arms: Exercise plus dietary intervention

SUMMARY:
Type 2 diabetes is a chronic disease that affects approximately 13% of Portuguese population and is associated with a high cardiovascular mortality by coronary artery disease and cerebrovascular disease and with a serious decline on well-being. Lifestyle changes are widely recommended to the control of type 2 diabetes and its complications. This study aims to analyse the effects of different community-based lifestyle programs (exercise or exercise plus dietary intervention) on health and well-being in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosed type 2 diabetes at least for six months;
2. Both genders;
3. Aged between 50 and 80 years old;
4. Non-smokers;
5. Not engaged in supervised exercise;
6. Community-dwelling;
7. Medical recommendation for lifestyle intervention;
8. Known medical history;
9. Diabetes complications under medical control (poor metabolic control, diabetic foot, diabetic retinopathy, diabetic nephropathy and diabetic autonomic neuropathy;
10. No cardiovascular, respiratory and musculoskeletal contraindications to exercise;
11. No gait and balance problems;
12. Not taking insulin or sulfonylureas for less than three months;
13. Volunteer participation with signed informed consent.

Exclusion Criteria:

1. Participation in another supervised exercise program during the study;
2. Participation in another supervised dietary intervention during the study;
3. Aggravation of a diabetes complication or another major health problem;

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Risk | Baseline, 9 and 21 months
  UKPDS Risk Engine
Health-Related Quality of Life | Baseline, 9 and 21 months
  SF-36 Health Survey

SECONDARY OUTCOMES:
Food Literacy | Baseline, 9 and 21 months
  General Nutrition Knowledge Questionnaire for Adults
Dietary Pattern | Baseline, 9 and 21 months
  3-day Food Record
Physical Fitness | Baseline, 9 and 21 months
  Physical Fitness Test Battery
Diabetic Foot Risk | Baseline, 9 and 21 months
  International Working Group on the Diabetic Foot Risk Classification)
Exercise-Related Adverse Events | Baseline, 9 and 21 months
  Number of acute injuries or adverse events during exercise sessions
Systolic Blood Pressure | Baseline, 9 and 21 months
  mmHg
Diastolic Blood Pressure | Baseline, 9 and 21 months
  mmHg
Glycemic Control | Baseline, 9 and 21 months
  Glycated Hemoglobin
Fast blood glucose | Baseline, 9 and 21 months
  mg/dL
Total Cholesterol | Baseline, 9 and 21 months
  mg/dL
Body Fat Mass | Baseline, 9 and 21 months
  Bioelectrical impedance analysis
Body Lean Mass | Baseline, 9 and 21 months
  Bioelectrical impedance analysis
Quality of Sleep | Baseline, 9 and 21 months
  Pittsburgh Sleep Quality Index
Symptoms of Anxiety and Depression | Baseline, 9 and 21 months
  Hospital Anxiety and Depression Scale
Chronic Pain | Baseline, 9 and 21 months
  Brief Pain Inventory Questionnaire
Diabetes-Dependent Quality of Life | Baseline, 9 and 21 months
  Audit of Diabetes-Dependent Quality of Life Questionnaire
Habitual Physical Activity | Baseline, 9 and 21 months
  International Physical Activity Questionnaire
Waist Circumference | Baseline, 9 and 21 months
  cm
Falls Risk | Baseline, 9 and 21 months
  Timed Up and Go Test
Sitting-Time | Baseline, 9 and 21 months
  Hours per day
Energy Expenditure | Baseline, 9 and 21 months
  kcal/kg/min
Body Mass Index | Baseline, 9 and 21 months
  kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Romeu Mendes, MD PhD, Principal Investigator — University of Trás-os-Montes e Alto Douro
Locations (1):
- University of Trás-os-Montes e Alto Douro, Vila Real, Portugal

REFERENCES:
- [Background] Matos M, Mendes R, Silva AB, Sousa N. Physical activity and exercise on diabetic foot related outcomes: A systematic review. Diabetes Res Clin Pract. 2018 May;139:81-90. doi: 10.1016/j.diabres.2018.02.020. Epub 2018 Feb 23. PMID 29477503
- [Result] Vasconcelos C, Almeida A, Cabral M, Ramos E, Mendes R. The Impact of a Community-Based Food Education Program on Nutrition-Related Knowledge in Middle-Aged and Older Patients with Type 2 Diabetes: Results of a Pilot Randomized Controlled Trial. Int J Environ Res Public Health. 2019 Jul 6;16(13):2403. doi: 10.3390/ijerph16132403. PMID 31284568
- [Result] Vasconcelos C, Almeida A, Sa C, Viana J, Cabral M, Ramos E, Mendes R. Nutrition-related knowledge and its determinants in middle-aged and older patients with type 2 diabetes. Prim Care Diabetes. 2020 Apr;14(2):119-125. doi: 10.1016/j.pcd.2019.06.007. Epub 2019 Jul 24. PMID 31350159
- See also: Official site — http://www.diabetesemmovimento.com